CLINICAL TRIAL: NCT05961176
Title: Exploratory Study on Bio-Signal Telemonitoring Using Electronic Textiles in a Pediatric Acute and Critical Care Setting
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Myant Medical Corp. (Industry)
Responsible Party: Principal Investigator, Aamir Jeewa, Staff Cardiologist, The Hospital for Sick Children
Other Study IDs: 1000079180
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
Keywords: Wearable Electronic Device; Cardiovascular Disease; Critical Care; Pediatric
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants and Children Admitted to the CCCU at SickKids: Inclusion Criteria: Patients from 1 month of age to 12 years of age who are admitted to SickKids CCCU with expected stays in CCCU longer than 12 hours including those for medical management and post-surgical patients.
  Interventions: Device: Skiin pediatric band and Skiin biometric pod

INTERVENTIONS:
Device: Skiin pediatric band and Skiin biometric pod — Infants that meet the inclusion criteria will be equipped with a Skiin pediatric band appropriate for their chest size. Heart rate, respiratory rate, temperature, and electrocardiogram will be monitored from 2 to 12 hours through the Skiin pediatric band and a standard of care device (Phillips Intellivue MX750) commonly used in the CCCU at SickKids.

SUMMARY:
The primary research objective is to determine the safety, feasibility, usability and validity of textile-enabled monitoring systems designed to capture physiologic variables, or "biological signals," related to cardiopulmonary function in children through comparison to hospital-based, standard-of-care monitoring in the Sickkids Cardiac Critical Care Unit (CCCU).

DETAILED DESCRIPTION:
This single-arm, non-randomized study is a usability, technology feasibility and data correlation study which will employ a convenience sampling method. The study will compare the quality of data obtained by the Myant Inc Skiin Pediatric Band smart textile device to the gold-standard data generated by the clinical devices in the CCCU at SickKids.

The primary research objective is to determine the safety, feasibility, usability and validity of textile-enabled monitoring systems designed to capture physiologic variables, or "biological signals," related to cardiopulmonary function in children through comparison to hospital-based, standard-of-care monitoring in the SickKids CCCU.

The secondary objectives are as follows; (1) To design textiles for infants and children that allow safe, developmentally appropriate care, (2) To investigate the optimum placement of biosensors to measure physiologic parameters such as heart and respiratory rate within the textile-based approach, (3) To validate the textile-based approach, including the integrated sensors, through comparison to physiologic data gathered as part of routine patient care through traditional comparative analysis, (4) To investigate usability of the textiles, including placement, removal, and effects on patient care activities, and (5) To gather clinician feedback on the textile use and design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from 1 month of age to 12 years of age who are admitted to SickKids CCCU with expected stays in CCCU longer than 12 hours including those for medical management and post-surgical patients.

Exclusion Criteria:

1. Any existing condition, diagnosis or physiologic state, in the opinion of the principal investigator, Co-Investigators or most responsible physicians, in which presence of the study monitoring system may have negative effects on patient status or may impair care delivered by the treating team (e.g. hemodynamic instability, at risk for acute deterioration in condition).
2. Patients with active wounds or devices (such as a chest tube or invasive lines) in areas that prohibit placement of all configurations of textile device. *
3. Patients with Methicillin-Resistant Staphylococcus aureus (MRSA) that represent an infection control risk.
4. Patients cannulated to extracorporeal membrane oxygenation (ECMO).
5. Patients with imaging/procedures scheduled outside of the CCCU within the 12 hours following eligibility assessment. **
6. Patients with an implanted cardioverter defibrillator (ICD)
7. Patients with a pacemaker, either implanted or temporary (temporary pacing wires not in use are allowed). ***
8. Patients whose chest/abdomen size is too large or small to fit the available sizes of the Skiin Pediatric Band.

Eligibility may be reassessed once an appropriate body location for the textile placement becomes available.*

Eligibility may be reassessed after the patient returns to the CCCU.**

Eligibility may be reassessed after the temporary pacemaker has been removed.***

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and Children Admitted to the Cardiac Critical Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-01-17 (Estimated); Study Completion 2026-01-17 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | collection during the single study session of 2-12 hours.
  The difference between heart rate measured from Skiin data and from standard of care device.
Respiratory Rate | collection during the single study session of 2-12 hours.
  The difference between respiratory rate measured from Skiin data and from standard of care device.
Temperature | collection during the single study session of 2-12 hours.
  The difference between temperature measured from Skiin data and from standard of care device.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Jeewa, MD, Principal Investigator — The Hospital for Sick Children; Michael-Alice Moga, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews RE, Fenton MJ, Ridout DA, Burch M; British Congenital Cardiac Association. New-onset heart failure due to heart muscle disease in childhood: a prospective study in the United kingdom and Ireland. Circulation. 2008 Jan 1;117(1):79-84. doi: 10.1161/CIRCULATIONAHA.106.671735. Epub 2007 Dec 17. PMID 18086928
- [Background] Wilkinson JD, Landy DC, Colan SD, Towbin JA, Sleeper LA, Orav EJ, Cox GF, Canter CE, Hsu DT, Webber SA, Lipshultz SE. The pediatric cardiomyopathy registry and heart failure: key results from the first 15 years. Heart Fail Clin. 2010 Oct;6(4):401-13, vii. doi: 10.1016/j.hfc.2010.05.002. PMID 20869642
- [Background] Kay JD, Colan SD, Graham TP Jr. Congestive heart failure in pediatric patients. Am Heart J. 2001 Nov;142(5):923-8. doi: 10.1067/mhj.2001.119423. No abstract available. PMID 11685182
- [Background] Nandi D, Rossano JW. Epidemiology and cost of heart failure in children. Cardiol Young. 2015 Dec;25(8):1460-8. doi: 10.1017/S1047951115002280. PMID 26675591
- [Background] Jacob E, Duran J, Stinson J, Lewis MA, Zeltzer L. Remote monitoring of pain and symptoms using wireless technology in children and adolescents with sickle cell disease. J Am Assoc Nurse Pract. 2013 Jan;25(1):42-54. doi: 10.1111/j.1745-7599.2012.00754.x. Epub 2012 Jul 12. PMID 23279278
- [Background] Zartner P, Handke R, Photiadis J, Brecher AM, Schneider MB. Performance of an autonomous telemonitoring system in children and young adults with congenital heart diseases. Pacing Clin Electrophysiol. 2008 Oct;31(10):1291-9. doi: 10.1111/j.1540-8159.2008.01180.x. PMID 18811810
- [Background] Zartner PA, Toussaint-Goetz N, Photiadis J, Wiebe W, Schneider MB. Telemonitoring with implantable electronic devices in young patients with congenital heart diseases. Europace. 2012 Jul;14(7):1030-7. doi: 10.1093/europace/eur434. Epub 2012 Feb 2. PMID 22308087
- [Background] Ware P, Ross HJ, Cafazzo JA, Laporte A, Seto E. Implementation and Evaluation of a Smartphone-Based Telemonitoring Program for Patients With Heart Failure: Mixed-Methods Study Protocol. JMIR Res Protoc. 2018 May 3;7(5):e121. doi: 10.2196/resprot.9911. PMID 29724704